CLINICAL TRIAL: NCT04263363
Title: A Prospective Digital Quality Improvement Project to Apply Best Clinical Practices to Patients at High Risk of Respiratory Complications
Brief Title: Applying Best Clinical Practices to Patients at High Risk of Respiratory Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Eilon Gabel, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Anes-Respiratory Dysfunction
Record Dates: First submitted 2020-01-17; First posted 2020-02-10 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Complication; Obstructive Sleep Apnea
Keywords: Respiratory Complication; Clinical Decision Support; Sugammadex
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: Historical prospective comparative effectiveness clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CDS pathway (Experimental): When the anesthesiologist completes the preoperative evaluation for a patient who is flagged as having either respiratory disease or OSA and will receive general anesthesia, the anesthesiologist will receive a pop-up window reminding them of the best practice guidelines for pulmonary management in high-risk patients. We anticipate that the pathway will suggest 1) use of sugammadex to reverse neuromuscular blockade if rocuronium was used 2) use of objective train of four monitoring throughout the case and to confirm reversal 3) use of a tidal volume of 6-8 cc/kg 4) use of at least 5 cmH2O of PEEP
  Interventions: Drug: Sugammadex 100 MG/ML [Bridion]

INTERVENTIONS:
Drug: Sugammadex 100 MG/ML [Bridion] — Sugammadex administered to patients within the clinical best practice pathway.
  Other Names: Bridion

SUMMARY:
The purpose of this study is to:

1. Perform a retrospective analysis on data contained in the UCLA Perioperative Data Warehouse on the incidence of respiratory dysfunction in the post-operative care unit (PACU) before and after the introduction of sugammadex into clinical practice.
2. Develop and implement a clinical best practice pathway designed to prevent postoperative respiratory complications in higher risk patients (such as those with OSA or preexisting respiratory disease) using education and clinical decision support in patients.

DETAILED DESCRIPTION:
This will be a historical prospective comparative effectiveness clinical trial where the investigators plan to leverage their experience in extracting data from the EMR as well as creating robust CDS pathways in order to create and implement a pathway to promote use of best respiratory care in patients receiving general anesthesia who are at increased risk for postoperative respiratory dysfunction. The overall study will consist of two parts:

1. Retrospective data analysis: The investigators will utilize the Perioperative Data Warehouse, a custom-built data warehouse, to study the effect of the introduction of sugammadex, a direct reversal agent for rocuronium, into clinical practice on time to "fitness for discharge" from the recovery room, as noted by the time the anesthesiologist places the discharge order, before and after intervention and postoperative respiratory dysfunction (as defined as duration of oxygen saturation below 90% in the PACU).
2. Creation and implementation of a pathway to prevent postoperative respiratory dysfunction: The investigators will design and implement a perioperative decision support system which will identify high-risk patients and provide best practice recommendations via electronic clinical decision support reminders.

Creation and implementation of a pathway to prevent postoperative respiratory dysfunction:

In order to improve outcomes for high-risk patients who receive general anesthesia and paralysis the investigators will design and implement a perioperative decision support system which will identify high-risk patients and provide best practice recommendations via electronic clinical decision support reminders. While the exact parameters of the pathway will be designed based upon feedback from a group of quality leaders in the department, in general the pathway will function as follows:

When the anesthesiologist completes the preoperative evaluation for a patient who is flagged as having either respiratory disease or OSA and will receive general anesthesia, the anesthesiologist will receive an alert reminding them of the best practice guidelines for pulmonary management in high-risk patients. As part of the study roll-out the investigators will present these guidelines with their quality committee, but anticipate that they will suggest 1) use of sugammadex to reverse neuromuscular blockade if rocuronium was used 2) use of objective train of four monitoring throughout the case and to confirm reversal 3) use of a tidal volume of 6-8 cc/kg 4) use of at least 5 cmH2O of PEEP.

The investigators anticipate running the prospective portion of the study for a one year data collection period. Specifically, they will allow a one month "wash out" period for pathway go live, followed by one year of data collection during which the pathway is live.

STUDY PROCEDURES

Pathway Design

The design of the pathway will undergo a well-established process that is designed to ensure buy-in and support from a large variety of providers within the Department of Anesthesiology and Perioperative Medicine at UCLA. The investigators will create a core group of individuals who represent key stakeholders in quality, informatics, and clinical decision making throughout our department. This group will be in charge of reviewing the existing literature and creating the pathway guidelines and associated decision support. The decision support will consist of preoperative alerts for high risk patients, intraoperative reminders for events such as ventilator settings and reversal as well as postoperative feedback on performance of identified best practices and outcomes. This pathway will include the recommendation of the use of sugammadex to reverse neuromuscular blockade and use of objective train of four (TOF) monitoring in high-risk individuals.

This core group will then present the recommended pathway for approval to our quarterly Quality Council and then broader Faculty Meetings for approval. The investigators estimate that the total time for pathway design and creation will be approximately 6 months.

Pathway Implementation

After approval, the investigators will work with the EMR build team in order to ensure the necessary modification to the EMR. After the modifications are complete, the investigators will establish a "go-live" date. After an initial period during which the investigators will accommodate feedback and ensure that the modifications were made successfully, no further modifications to the respiratory pathway will be made. The investigators plan to keep this pathway in place for at least one year (the study period).

Data Collection and Analysis

As noted above, the team has the ability to automatically collect the data from the EMR for analysis purposes. After the one year implementation period investigators will extract the data elements noted above for the study period as well as an equivalent period prior to pathway implementation. The data will be analyzed for the overall application of best practices before and after as well as a change in primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* UCLA Ronald Reagan or Santa Monica patients aged 18 and older who had a general anesthetic with either rocuronium or vecuronium.
* Patients who receive sugammadex from the specified study supply

Exclusion Criteria:

* Patients under the age of 18
* Patients with a preoperative glomerular filtration rate less than 30 or on hemodialysis
* Patients with known hypersensitivity to any of the following: rocuronium, vecuronium, sugammadex, neostigmine or glycopyrrolate
* Patients with known neuromuscular disease
* Patients who remain intubated after surgery or leave the operating room with a tracheostomy in-situ
* Patients who did not receive reversal of neuromuscular blockade (with neostigmine in the pre-period or sugammadex in the post-period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12248 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-Trial Cohort Timeframe: Patients from 2015, before sugammadex was available on the market (pre-2016).
  Purpose: Served as a historical control group to compare outcomes before the introduction of sugammadex.
  Size: 6,824 patients. Post-Trial Cohort Timeframe: Patients enrolled between February 2022 and May 2024. Purpose: Identified and enrolled via an automated system using Best Practice Advisories (BPAs) in the EHR.
  Size: 5,424
Period: Pre-Trial Cohort
Arm/Group | CDS Pathway
Started | 6824
Completed | 6824
Not Completed | 0
Period: Post-Trial Cohort
Arm/Group | CDS Pathway
Started | 5424
Completed | 5424
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pre-Trial Cohort
  * Timeframe: Patients from 2015, before sugammadex was available on the market (pre-2016).
  * Purpose: Served as a historical control group to compare outcomes before the introduction of sugammadex.
  * Size: 6,824 patients.
  Post-Trial Cohort
  * Timeframe: Patients enrolled between February 2022 and May 2024.
  * Purpose: Identified and enrolled via an automated system using Best Practice Advisories (BPAs) in the EHR.
  * Size: 5,424
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12,248
Age, Customized [Count of Participants; unit: Participants]
  ≥18 | 12248
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Pre-Trial Cohort: Size: 6,824 patients.
  Post-Trial Cohort: Size: 5,424 patients.
  Participants
    Pre-Trial Sex: number analyzed (Participants) | 6824
    Pre-Trial Sex: Male | 3249
    Pre-Trial Sex: Female | 3575
    Pre-Trial Sex: Unknown | 0
    Post-Trial Sex: number analyzed (Participants) | 5424
    Post-Trial Sex: Male | 2525
    Post-Trial Sex: Female | 2897
    Post-Trial Sex: Unknown | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Pre-Trial Cohort: Size: 6,824 patients.
  Post-Trial Cohort: Size: 5,424 patients.
  Participants
    Pre-Trial Race: number analyzed (Participants) | 6824
    Pre-Trial Race: American Indian or Alaska Native | 36
    Pre-Trial Race: Asian | 605
    Pre-Trial Race: Black or African American | 578
    Pre-Trial Race: Middle Eastern/North African | 34
    Pre-Trial Race: Native Hawaiian or Other Pacific Islander | 37
    Pre-Trial Race: Unknown / Not Specified | 1198
    Pre-Trial Race: White | 4336
    Post-Trial Race: number analyzed (Participants) | 5424
    Post-Trial Race: American Indian or Alaska Native | 62
    Post-Trial Race: Asian | 504
    Post-Trial Race: Black or African American | 379
    Post-Trial Race: Middle Eastern/North African | 119
    Post-Trial Race: Native Hawaiian or Other Pacific Islander | 29
    Post-Trial Race: Unknown / Not Specified | 1142
    Post-Trial Race: White | 3189
Region of Enrollment [Number; unit: participants]
  United States | 12248

OUTCOME MEASURES:

1. Primary Outcome: Time to "Fitness for Discharge" From the Recovery Room
Description: The time the anesthesiologist places the discharge order
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Pre-Trial 6,824. Post-Trial 5,424.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12,248
Minutes
  Pre-Trial: number analyzed (Participants) | 6824
  Pre-Trial | 165.64 (89.69)
  Post-Trial: number analyzed (Participants) | 5424
  Post-Trial | 154.60 (86.17)

2. Primary Outcome: Incidence of Hypoxemia in the PACU (Oxygen Saturation Below 90%)
Description: Documentation oxygen saturation below 90%
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Pre-Trial 6,824. Post-Trial 5,424.
Measure: Count of Participants; unit: Participants
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12,248
Participants
  Pre-Trial | 18
  Post-Trial | 9
  No Incidence | 12,221

3. Secondary Outcome: Percentage of Patients Who Had Intraoperative Lung Protective Ventilation
Description: Percentage of patients who had intraoperative lung protective ventilation prior to extubation
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: This outcome was not measured due to impacted hospital regulations during COVID-19. Hospital regulations restricted this measurement to be taken as intake volume was low and therefore hospital administration deemed it uncollectable at the time. Therefore, this measurement was never completed during the duration of the study as our team were required to follow updated hospital regulations.
Arm/Group | CDS Pathway
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Hypoxemia in the PACU (Oxygen Saturation Below 95%)
Description: Documentation of oxygen saturation below 95%
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Pre-Trial 6,824. Post-Trial 5,424.
Measure: Count of Participants; unit: Participants
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12,248
Participants
  Pre-Trial | 421
  Post-Trial | 1170
  No Incidence | 10,657

5. Secondary Outcome: Duration of Supplemental Oxygen Needed by High-risk Patients
Description: Duration of supplemental oxygen needed by high-risk patients before and after intervention
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: as for outcome 3
Arm/Group | CDS Pathway
Number analyzed (Participants) | 0

6. Secondary Outcome: Postoperative Reintubation Rate
Description: Rate of postoperative reintubation
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Analysis was completed for Post-Trial participants equaling 5,424.
Measure: Count of Participants; unit: Participants
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12248
Participants
  Pre-Trial: number analyzed (Participants) | 6824
  Pre-Trial | 13
  Post-Trial: number analyzed (Participants) | 5424
  Post-Trial | 4

7. Secondary Outcome: Number of Patients With Unplanned Upgrade of Care
Description: Number of patients with unplanned upgrade of care
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Pre-Trial 6,824. Post-Trial 5,424.
Measure: Count of Participants; unit: Participants
Arm/Group | CDS Pathway
Number analyzed (Participants) | 12248
Participants
  Pre-Trial | 128
  Post-Trial | 16
  No Incidence | 12,104

8. Secondary Outcome: Percentage of Patients Who Had Train of Four Ratio Measurement
Description: Percentage of patients who had Train of Four ratio measurement prior to extubation
Time Frame: One year prior to study intervention to one year following implementation of study intervention
Population: Analysis was only completed for Post-Trial participants equaling 5,424. Analysis could not be collected for Pre-Trial group as the Pre-Trial group was collected retrospectively and this measurement was not implemented into care until the prospective collection of the Post-Trial group. Therefore, we could not obtain the Pre-Trial group's measurements as these measurements had never been collected to obtain retrospectively.
Measure: Count of Participants; unit: Participants
Arm/Group | CDS Pathway
Number analyzed (Participants) | 5424
Participants | 2704

ADVERSE EVENTS:
Time Frame: Time of consent up to 48 hours post drug administration.
Description: AEs collected for bradycardia, anaphylaxis, and reintubation cases.
Groups:
- CDS Pathway (Pre-Trial); CDS Pathway (Post-Trial): When the anesthesiologist completes the preoperative evaluation for a patient who is flagged as having either respiratory disease or OSA and will receive general anesthesia, the anesthesiologist will receive a pop-up window reminding them of the best practice guidelines for pulmonary management in high-risk patients. We anticipate that the pathway will suggest 1) use of sugammadex to reverse neuromuscular blockade if rocuronium was used 2) use of objective train of four monitoring throughout the case and to confirm reversal 3) use of a tidal volume of 6-8 cc/kg 4) use of at least 5 cmH2O of PEEP
  Sugammadex 100 MG/ML [Bridion]: Sugammadex administered to patients within the clinical best practice pathway.
Arm/Group | CDS Pathway (Pre-Trial) | CDS Pathway (Post-Trial)
All-Cause Mortality (participants affected / at risk) | 0/6824 | 0/5424
Serious Adverse Events (participants affected / at risk) | 0/6824 | 8/5424
Other Adverse Events (participants affected / at risk) | 0/6824 | 0/5424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDS Pathway (Pre-Trial) (N=6824) | CDS Pathway (Post-Trial) (N=5424)
Bradycardia (Cardiac disorders) | 0 (0) | 4 (4)
Anaphylaxis (Immune system disorders) | 0 (0) | 2 (2)
Reintubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT04263363/Prot_SAP_000.pdf